CLINICAL TRIAL: NCT05505136
Title: Mobile Cardiac Telemetry and Advanced Multi-Parameter Monitoring in PatientS Wearing a Novel Device With Biometric Based
Brief Title: Mobile Cardiac Telemetry and Advanced Multi-Parameter Monitoring in PatientS Wearing a Novel Device With Biometric Based Medications Changes
Acronym: MAPS II
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0255
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MAPS Study Patients with Medication Change Reported: No intervention will be administered. This is a retrospective study of the patients who participating in the MAPS Protocol 90D0234 completed in 2021. Patients who had a medication change reported in that study are the focus of this study MAPS II 90D0255.
  Interventions: Device: Arrhythmia Management System (AMS)

INTERVENTIONS:
Device: Arrhythmia Management System (AMS) — Retrospective collection of data related to subjects who participated in the MAPS 90D0234 study and had a medication change reported will wearing the AMS device.

SUMMARY:
To determine the associations among biometric data and previously reported medication changes in the original MAPS study

DETAILED DESCRIPTION:
1. Each center that previously reported making a medication change in a MAPS patient based on biometric information will complete a case report form detailing the rhythm, symptom, medication and dosage change, and which biometric(s) were used to make this decision.
2. Follow up at 6 months will be determined for all patients to assess the impact of the medication change.

ELIGIBILITY:
Inclusion Criteria:

* those that completed the MAPS study and that had medication changes based wholly or in part on biometric information.

Exclusion Criteria:

* Those patients from the MAPS study that did not have medication changes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who completed the MAPS study with a reported medication change based wholly or in part on biometric information.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Association Between Arrhythmia Biometric and Medication Change | 1 Day
  Clinical Case Report Form
Association Between Subject-Reported Symptom Biometric and Medication Change | 1 Day
  Clinical Case Report Form
Association Between Subject Wellness Biometric and Medication Change | 1 Day
  Clinical Case Report Form
Association Between Subject Adverse Event and Medication Change | 1 Day
  Clinical Case Report Form
Association Between Subject Status and Medication Change | 1 Day
  Clinical Case Report Form
Association Between Subject Hospital Events and Medication Change | 1 Day
  Clinical Case Report Form
Association Between Subject Clinical Events and Medication Change | 1 Day
  Clinical Case Report Form

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ringquist, Study Chair — Zoll Services LLC
Locations (8):
- United States (8):
  - Cardiovascular Institute of Central Florida, Ocala, Florida
  - First Coast Heart & Vascular Center, Saint Augustine, Florida
  - Jackson Heart Clinic, Jackson, Mississippi
  - PharmaTex Research, Amarillo, Texas
  - Texas Cardiology Associates of Houston, Kingwood, Texas
  - CardioVoyage, McKinney, Texas
  - Dr. Daniel W. Gottlieb, Burien, Washington
  - St. Mary's Medical Center EP, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No